CLINICAL TRIAL: NCT01710150
Title: Randomized Trial Comparing Long Term Occurrence of Atrial Arrhythmias Including Atrial Fibrillation (AF) and Thromboembolic Complications in Patients With Typical Atrial Flutter (AFLT) Undergoing Cavo-tricuspid Isthmus (CTI) Ablation Alone Versus CTI Ablation Combined With Pulmonary Vein Isolation (PVI).
Brief Title: Pulmonary Vein Isolation To Reduce Future Risk Of Atrial Fibrillation In Patients Undergoing Typical Flutter
Acronym: REDUCE AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REDUCE AF
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Typical Atrial Flutter; Risk Factors With Future Development of Atrial Flutter
Keywords: typical aflutter (AFLT); CTI ablation; Atrial Fibrillation (AF); PVI
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTI ablation only (Placebo Comparator): subjects undergoing cavo-tricuspid isthmus (CTI) ablation alone for Atrial flutter
  Interventions: Procedure: CTI ablation alone
- CTI ablation and PVI. (Active Comparator): subjects undergoing cavo-tricuspid isthmus (CTI) ablation for Atrial flutter and pulmonary vein isolation (PVI) for Atrial Fibrillation.
  Interventions: Procedure: CTI ablation and Pulmonary vein isolation (PVI)

INTERVENTIONS:
Procedure: CTI ablation alone
  Arms: CTI ablation only
Procedure: CTI ablation and Pulmonary vein isolation (PVI)
  Arms: CTI ablation and PVI.

SUMMARY:
The purpose is to compare long term occurrence of atrial arrhythmias including atrial fibrillation (AF) and thromboembolic complications including cerebrovascular events (CVE) in patients with typical atrial flutter (AFLT) undergoing cavo-tricuspid isthmus (CTI) ablation alone versus CTI ablation combined with pulmonary vein isolation (PVI).

DETAILED DESCRIPTION:
Typical Atrial Flutter (AFLT) is a common cardiac arrhythmia. Studies have demonstrated the safety and superiority of ablation procedure over antiarrhythmic drug (AAD) therapy. Long term freedom from typical AFLT has been consistently shown after successful ablation, but up to 30% of these patients can experience new onset of a different arrhythmia i.e., Atrial Fibrillation (AF). AF results from triggers in the back of the left upper chamber in the heart (left atrium - LA). These triggers typically arise from in and around the opening of the 4 veins (pulmonary veins - PVs) that bring blood from the lungs into the heart. The highest incidence of AF in patients undergoing ablation for typical AFLT was observed where the follow-up duration exceeded a year after the AFLT ablation. This would suggest that AF development in patients undergoing typical AFLT ablation is progressive and inevitable.

ELIGIBILITY:
Inclusion Criteria:

All patients with typical AFLT confirmed by a 12-lead ECG that are referred for ablation and manifest ≥ 2 risk factors associated with future development of AF will be eligible to participate in the study.

Risk factors for predicting future occurrence of AF will include:

1. prior remote history of AF (≤ 2 episodes ≥ 1 year from the date of evaluation for study participation),
2. LA size > 4.0 cm,
3. left ventricular ejection fraction (LVEF) ≤ 50%,
4. hypertension, and/or 5) obstructive sleep apnea.

Exclusion Criteria:

1. Subjects with documented ≥ 2 AF episodes within the preceding 6 months of enrollment,
2. inability or unwillingness to take 6 weeks of oral anticoagulation after the procedure and
3. failure to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Primary: 1) Long-term (~2 year) freedom from atrial arrhythmias (AFLT and / or AF) and thromboembolic events (including CVEs). | 2 years

SECONDARY OUTCOMES:
Occurrence of serious adverse events [CVE, pericardial effusion results in tamponade, development of PV stenosis (symptomatic or asymptomatic >70% reduction in PV diameter in ≥1 veins assessed by CT scan), left atrial-esophageal fistula and death | 2 years

OTHER OUTCOMES:
Long term (~2 year) use of membrane stabilizing antiarrhythmic drugs. Long term (~2 year) use of oral anticoagulation. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Dixit, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mohanty S, Natale A, Mohanty P, DI Biase L, Trivedi C, Santangeli P, Bai R, Burkhardt JD, Gallinghouse GJ, Horton R, Sanchez JE, Hranitzky PM, Al-Ahmad A, Hao S, Hongo R, Beheiry S, Pelargonio G, Forleo G, Rossillo A, Themistoclakis S, Casella M, Russo AD, Tondo C, Dixit S. Pulmonary Vein Isolation to Reduce Future Risk of Atrial Fibrillation in Patients Undergoing Typical Flutter Ablation: Results from a Randomized Pilot Study (REDUCE AF). J Cardiovasc Electrophysiol. 2015 Aug;26(8):819-825. doi: 10.1111/jce.12688. Epub 2015 May 26. PMID 25884325